CLINICAL TRIAL: NCT02850536
Title: Phase Ib Trial of CAR-T Hepatic Artery Infusions or Pancreatic Venous Infusions Delivered With the Surefire Infusion System (SIS) for CEA-Expressing Liver Metastases or Pancreas Cancer
Brief Title: CAR-T Hepatic Artery Infusions or Pancreatic Venous Infusions for CEA-Expressing Liver Metastases or Pancreas Cancer
Acronym: HITM-SURE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Roger Williams Medical Center (Other)
Collaborators: University of Colorado, Denver (Other); Sorrento Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 350-74
Record Dates: First submitted 2016-07-14; First posted 2016-08-01 (Estimated); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Liver Metastases
Keywords: Colorectal Cancer; Liver Metastases; Breast Cancer; Gastric Cancer; Pancreas Cancer; Carcinoembryonic antigen; CAR-T; Immunotherapy
MeSH Terms: conditions — Colorectal Neoplasms; Breast Neoplasms; Stomach Neoplasms; Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- anti-CEA CAR-T cells (Experimental): Three infusions of gene-modified anti-CEA T cells over the course of 3 weeks into the hepatic artery via a percutaneous approach along with low dose IL-2.
  Interventions: Biological: anti-CEA CAR-T cells

INTERVENTIONS:
Biological: anti-CEA CAR-T cells — Gene modified patient T cells
  Other Names: Designer T cells

SUMMARY:
This is an open label, fixed dose, phase Ib trial of anti-CEA CAR-T cell infusions delivered via the hepatic artery or splenic vein using the Surefire Infusion System (SIS) for patients with CEA-expressing liver metastases or pancreas cancer.

DETAILED DESCRIPTION:
Patients undergo leukapheresis from which peripheral blood mononuclear cells are purified. T cells are activated and then re-engineered to express chimeric antigen receptors (CARs) specific for CEA. Cells are expanded in culture and returned to the patient by percutaneous hepatic artery infusion at specific cell doses. Prior to the first dose, each patient will undergo diagnostic angiography to verify suitable arterial anatomy. Three anti-CEA CAR-T doses per patient are planned at 1-week intervals. Low dose interleukin-2 will be given via an ambulatory infusion pump for 4 weeks. Normal liver and tumor biopsies will be obtained at the time of the initial diagnostic angiogram and during the final session following the 3rd CAR-T infusion.

Patients with CEA+ liver metastases who exhibit in-liver control following CAR-T therapy who also have CEA+ primary pancreatic tumors may be eligible to receive direct intrapancreatic CAR-T retrograde venous infusions. A maximum of 2 infusions will be delivered. No additional IL-2 will be given and there will be no additional biopsies.

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically confirmed diagnosis of CEA+ adenocarcinoma and liver metastases. Patient must have either histologic confirmation of the liver metastases or histologic documentation of the primary tumor and definitive radiologic evidence of liver involvement. Measurable disease is required with lesions of > 1.0 cm by CT. Soluble CEA is not acceptable as the sole measure of disease. Limited extrahepatic disease is acceptable if confined to the lungs or peritoneal cavity.
* Tumor must be CEA-expressing as demonstrated by elevated serum CEA levels (≥10ng/ml) or immunohistochemistry on a biopsy specimen. Archived tissue is acceptable for determination of CEA expression.
* Patient must be at least 18 years of age.
* Patient able to understand and sign informed consent.
* Patient with a life expectancy of greater than four months.
* Patient failed at least one line of standard systemic chemotherapy and has unresectable disease.
* Patient with performance status of 0 to 1 (ECOG).
* Patient with adequate organ function as defined in protocol.
* Acceptable hepatic vascular anatomy as determined by CT, MR, or conventional angiography. A nuclear medicine study will be performed to document the absence of a significant hepatic-pulmonary shunt (<20%).

Exclusion Criteria:

* Female patients of childbearing age will be tested for pregnancy. Pregnant patients will be excluded from the study. Males who are actively seeking to have children will be made aware of the unknown risks of this study protocol on human sperm and the need to practice birth control.
* Patients with serious or unstable renal, hepatic, pulmonary, cardiovascular, endocrine, rheumatologic, or allergic disease based on history, physical exam and laboratory tests will be excluded, as outlined in section 5.2.8.
* Patients with active clinical disease caused by CMV, hepatitis B or C, HIV or tuberculosis will be excluded from the study.
* Patients who have had cytotoxic and/or radiation therapy within 4 weeks prior to entry into the trial or 4 weeks prior to infusion will be excluded. Patients with other concurrent malignancies will be excluded.
* Patients requiring systemic steroids will be excluded.
* Patients with unsuitable hepatic vascular anatomy will be excluded from the study.
* Patients with extrahepatic metastatic disease beyond the lungs or abdominal/ retroperitoneal lymph nodes.
* Patients with >50% liver replacement at time of treatment will be excluded.
* Previous external beam radiotherapy to the liver.
* Portal vein thrombosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2021-09-17 (Actual)

PRIMARY OUTCOMES:
Safety of CAR-T cell hepatic artery infusions delivered using the Surefire Infusion System (SIS) as Measured by Number of Participants with Adverse Events | 10 weeks
  To determine the safety and regimen limiting toxicity (RLT) of anti-CEA CAR-T hepatic artery infusions (HAI) via the Surefire Infusion System (SIS) for CEA-expressing liver metastases

SECONDARY OUTCOMES:
Radiographic treatment response by MRI | 10 weeks
  Changes in tumor size
Radiographic treatment response by PET | 10 weeks
  Changes in tumor metabolic activity
CAR-T detection in liver tumors | 10 weeks
  Quantification of CAR-T cells in liver tumor core biopsies
CAR-T detection in normal liver tissue | 10 weeks
  Quantification of CAR-T cells in normal liver core biopsies
CAR-T detection in extrahepatic sites | 10 weeks
  Quantification of CAR-T in blood samples
Serum Cytokine Levels | 10 weeks
  Measurement of cytokines as indicators of immune response
CEA level | 10 weeks
  Measurement of serum tumor marker (ng/ml)
Tumor biopsy | 10 weeks
  Assessment of tumor necrosis and fibrosis
Safety of Direct Intrapancreatic CAR-T Retrograde Venous Infusions (RVI) Delivered Using the Surefire Infusion System (SIS) | 10 weeks
  RVI via the Surefire Infusion System (SIS) for CEA+ Primary Pancreatic Tumors Following In-liver Disease Control

CONTACTS AND LOCATIONS:
Overall Officials: Steven C. Katz, MD, Principal Investigator — Roger Williams Medical Center; Richard Schulick, MD, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Hospital, Aurora, Colorado
  - Roger Williams Medical Center, Providence, Rhode Island

REFERENCES:
- [Derived] Katz SC, Moody AE, Guha P, Hardaway JC, Prince E, LaPorte J, Stancu M, Slansky JE, Jordan KR, Schulick RD, Knight R, Saied A, Armenio V, Junghans RP. HITM-SURE: Hepatic immunotherapy for metastases phase Ib anti-CEA CAR-T study utilizing pressure enabled drug delivery. J Immunother Cancer. 2020 Aug;8(2):e001097. doi: 10.1136/jitc-2020-001097. PMID 32843493